CLINICAL TRIAL: NCT01115192
Title: Blephacura Versus Baby Shampoo to Treat Blepharitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Optima Pharmazeutische GmbH (Unknown)
Responsible Party: Principal Investigator, Arno Hueber, Blephacura Versus Baby Shampoo to Treat Blepharitis, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OptimaCologne
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients with chronic blepharitis, that will be treated with blephacura
  Interventions: Procedure: Group A
- Group B (Experimental): Patients with chronic blepharitis that will be treated with diluted baby shampoo
  Interventions: Procedure: Group B

INTERVENTIONS:
Procedure: Group A — Blephacura is a solution with liposomes and used for cleaning of the eye lid to treat blepharitis
  Arms: Group A
Procedure: Group B — Diluted Baby Shampoo is used for cleaning of the eye lid to treat blepharitis
  Arms: Group B

SUMMARY:
The aim of the study is to compare the effectiveness in treatment of chronic blepharitis either with a phospholipid liposome suspension compared to a conventional therapy recommendation using diluted baby shampoo.

ELIGIBILITY:
Inclusion Criteria:

* patients with blepharitis
* 100 eyes of 100 patients (50 patients treated with Blephacura, 50 patients treated with diluted baby shampoo) The ratio of female / male is not involved.

Exclusion Criteria:

* all patients that are not included in the group of inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, University of Cologne, Cologne, North Rhine-Westphalia, Germany